CLINICAL TRIAL: NCT05518747
Title: Effect of Probiotics as Supplement to Non-surgical Periodontal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Daniel Belstrøm, DDS, PhD, Associate professor, dr. odont., PhD, DDS, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCPH_01_007
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double blinded randomized clinical trial with a test and placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computerized randomization only known to the principal investigator, who are not directly involved in data collection or data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): In this group participants will receive non-surgical periodontal treatment at baseline, which will for 12 weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): In this group participants will receive non-surgical periodontal treatment at baseline, which will for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — In this group participants will receive probiotic supplements twice a day (morning and evening) for a period of 12 weeks.
  Arms: Probiotic
Dietary Supplement: Placebo — In this group participants will receive placebo twice a day (morning and evening) for at period of 12 weeks.
  Arms: Placebo

SUMMARY:
The present study is a double-blinded randomized clinical trial with a duration of 12 weeks.

DETAILED DESCRIPTION:
The present study is a double-blinded randomized clinical trial with a duration of 12 weeks

. 60 patients with periodontitis stage 2-3, grade B-C, generalized will be allocated in the test (probiotic) and the control (placebo) group at baseline.

The intervention is non-surgical periodontal treatment, which will be applied at baseline and followed for 12 weeks.

Clinical measurements and sampling will be performed at baseline, week 6 and week 12.

Primary endpoint: Changes in microbial composition.

Secondary endpoints: Changes in clinical and immunological parameters

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage 2-3, Grade B-C, generalized

Exclusion Criteria:

* • Use of systemic antibiotics within the latest three months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in microbial composition in dental plaque | Baseline vs. week 6 and week 12
  Changes in alpha and beta diversity of microbial composition

SECONDARY OUTCOMES:
Changes in dental plaque | Baseline vs. week 6 and week 12
  Changes in mean level of dental plaque
Changes in bleeding on probing | Baseline vs. week 6 and week 12
  Changes in mean level of bleeding on probing
Changes in probing pocket depth | Baseline vs. week 6 and week 12
  Changes in mean level of probing pocket depth
Changes in clinical attachment level | Baseline vs. week 6 and week 12
  Changes in mean level of clinical attachment level
Changes in salivary levels of inflammatory cytokines | Baseline vs. week 6 and week 12
  Changes in mean salivary levels of selected inflammatory cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Odontology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
All microbial data will be shared, as these will be uploaded to a publically accessible database.
  In accordance with GDPR, immunological and clinical data will only be shared as mean (range) values.